CLINICAL TRIAL: NCT04762511
Title: A Phase I, Single-blind, Randomised, Placebo-controlled, Dose Escalation Study to Evaluate the Reactogenicity, Safety and Immune Response of an HSV Vaccine in Healthy Participants Aged 18-40 Years
Brief Title: A Study on the Reactogenicity, Safety and Immune Response of a Vaccine Against Herpes Simplex Virus (HSV)-2 in Healthy Participants Aged 18-40 Years
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: To enable development of an enhanced version of the vaccine
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 213830
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Herpes Simplex
Keywords: First Time in Human; Vaccine; Healthy participants; Herpes Simplex Virus; Reactogenicity; Safety; Immune response
MeSH Terms: conditions — Herpes Simplex | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- HSV lower dose formulation Group (Experimental): Healthy participants, 18 to 40 years of age, receive two doses of the HSV lower dose formulation vaccine intramuscularly, one at Day 1 and one at Day 57.
  Interventions: Biological: Lower dose formulation of HSV vaccine (GSK4108771A)
- Placebo Step 1 Group (Placebo Comparator): Healthy participants, 18 to 40 years of age, receive two doses of placebo (saline) intramuscularly, one at Day 1 and one at Day 57.
  Interventions: Drug: Placebo (saline)
- HSV low dose formulation Group (Experimental): Healthy participants, 18 to 40 years of age, receive two doses of the HSV low dose formulation vaccine intramuscularly, one at Day 1 and one at Day 57.
  Interventions: Biological: Low dose formulation of HSV vaccine (GSK4108771A)
- Placebo Step 2 Group (Placebo Comparator): Healthy participants, 18 to 40 years of age, receive two doses of placebo (saline) intramuscularly, one at Day 1 and one at Day 57.
  Interventions: Drug: Placebo (saline)
- HSV medium dose formulation Group (Experimental): Healthy participants, 18 to 40 years of age, receive two doses of the HSV medium dose formulation vaccine intramuscularly, one at Day 1 and one at Day 57.
  Interventions: Biological: Medium dose formulation of HSV vaccine (GSK4108771A)
- Placebo Step 3 Group (Placebo Comparator): Healthy participants, 18 to 40 years of age, receive two doses of placebo (saline) intramuscularly, one at Day 1 and one at Day 57.
  Interventions: Drug: Placebo (saline)
- HSV high dose formulation Group (Experimental): Healthy participants, 18 to 40 years of age, receive two doses of the HSV high dose formulation vaccine intramuscularly, one at Day 1 and one at Day 57.
  Interventions: Biological: High dose formulation of HSV vaccine (GSK4108771A)
- Placebo Step 4 Group (Placebo Comparator): Healthy participants, 18 to 40 years of age, receive two doses of placebo (saline) intramuscularly, one at Day 1 and one at Day 57.
  Interventions: Drug: Placebo (saline)

INTERVENTIONS:
Biological: Lower dose formulation of HSV vaccine (GSK4108771A) — 2 doses of the lower dose formulation of HSV vaccine (GSK4108771A) administered intramuscularly in the non-dominant arm, one each at Day 1 and Day 57.
  Arms: HSV lower dose formulation Group
Biological: Low dose formulation of HSV vaccine (GSK4108771A) — 2 doses of the low dose formulation of HSV vaccine (GSK4108771A) administered intramuscularly in the non-dominant arm, one each at Day 1 and Day 57.
  Arms: HSV low dose formulation Group
Biological: Medium dose formulation of HSV vaccine (GSK4108771A) — 2 doses of the medium dose formulation of HSV vaccine (GSK4108771A) administered intramuscularly in the non-dominant arm, one each at Day 1 and Day 57.
  Arms: HSV medium dose formulation Group
Biological: High dose formulation of HSV vaccine (GSK4108771A) — 2 doses of the high dose formulation of the HSV vaccine (GSK4108771A) administered intramuscularly in the non-dominant arm, one each at Day 1 and Day 57.
  Arms: HSV high dose formulation Group
Drug: Placebo (saline) — 2 doses of placebo (saline) administered intramuscularly in the non-dominant arm, one each at Day 1 and Day 57.
  Arms: Placebo Step 1 Group; Placebo Step 2 Group; Placebo Step 3 Group; Placebo Step 4 Group

SUMMARY:
The purpose of this first-time-in-human (FTiH) study is to assess the reactogenicity, safety and immunogenicity of four different dose levels of an experimental herpes simplex virus type 2 (HSV-2) vaccine, when administered intramuscularly (IM) on a 0, 2-month schedule to healthy participants aged 18-40 years.

ELIGIBILITY:
Inclusion Criteria:

* Participants, who, in the opinion of the investigator, can and will comply with the requirements of the Protocol.
* Written informed consent obtained from the participant prior to performance of any study-specific procedure.
* Healthy participants as established by medical history and clinical examination before entering into the study.
* Man or woman aged 18-40 years, included, at the time of the first vaccination.
* Women of non-childbearing potential may be enrolled in the study.
* Women of childbearing potential may be enrolled in the study, if the participant:

  * Has practiced adequate contraception for one month prior to vaccination, and;
  * Has a negative pregnancy test result on the day of vaccination, and;
  * Has agreed to continue adequate contraception until the end of the study.
* Seronegative for HIV, as determined by laboratory screening tests. Participants documented to be positive to HIV will not be eligible for study participation.
* Seronegative for HSV-2 as determined by Western blot.

Exclusion Criteria:

Medical Conditions

* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study vaccines.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Hypersensitivity to latex.
* Acute or chronic clinically significant pulmonary, cardiovascular, hepatic, endocrine, or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Recurrent history or uncontrolled neurological disorders or seizures.
* Grade 2 or higher haematological and/or biochemical laboratory abnormality at screening.
* Body mass index ≤ 18 kg/m^2 or ≥ 35 kg/m^2.
* History of any form of ocular HSV infection, HSV-related erythema multiforme, or HSV-related neurological complications.
* Participants with symptoms suggestive of Coronavirus disease 2019 (COVID-19) infection within 14 days before the first study vaccination. Participants should be free of symptoms for at least 14 days.
* Participants with known COVID-19-positive contacts in the past 14 days before the first study vaccination.

Prior/Concomitant Therapy

* Use of any investigational or non-registered product other than the study vaccines during the period beginning 30 days before the first dose of study vaccine (Day -29 to Day 1), or planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the Protocol in the period starting 15 days before each dose and ending 15 days after each dose of study vaccine administration.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting three months before the first dose of study vaccine or planned administration during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting three months prior to the first study vaccine dose. For corticosteroids, this will mean prednisone equivalent ≥ 20 mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Prior receipt of another vaccine containing HSV-2 antigens. Prior/Concurrent Clinical Study Experience
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product.

Other Exclusions

* Pregnant or lactating woman.
* Woman planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Percentage of participants reporting solicited administration site events within 7 days after the first vaccine dose administered at Day 1 | Within 7 days after the first vaccine dose (administered at Day 1)
  The solicited administration site events are pain, redness and swelling.
Percentage of participants reporting solicited administration site events within 7 days after the second vaccine dose administered at Day 57 | Within 7 days after the second vaccine dose (administered at Day 57)
  The solicited administration site events are pain, redness and swelling.
Percentage of participants reporting solicited systemic events within 7 days after the first vaccine dose administered at Day 1 | Within 7 days after the first vaccine dose (administered at Day 1)
  The solicited systemic events are fever, fatigue, headache, nausea, vomiting, diarrhoea, abdominal pain, myalgia and arthralgia. The preferred location for measuring temperature is the oral cavity. Fever is defined as temperature equal to or above (≥) 38.0 degree Celsius (°C)/ 100.4°F, regardless the location of measurement.
Percentage of participants reporting solicited systemic events within 7 days after the second vaccine dose administered at Day 57 | Within 7 days after the second vaccine dose (administered at Day 57)
  The solicited systemic events are fever, fatigue, headache, nausea, vomiting, diarrhoea, abdominal pain, myalgia and arthralgia. The preferred location for measuring temperature is the oral cavity. Fever is defined as temperature equal to or above (≥) 38.0 degree Celsius (°C)/ 100.4°F, regardless the location of measurement.
Percentage of participants reporting unsolicited adverse events (AEs) within 28 days after the first vaccine dose administered at Day 1 | Within 28 days after the first vaccine dose (administered at Day 1)
  An unsolicited AE is any untoward medical occurrence (an unfavourable/unintended sign - including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant that is temporally associated with the study intervention, whether or not considered related to the study intervention and that was not included in a list of solicited events using a Participant Diary.
Percentage of participants reporting unsolicited adverse events (AEs) within 28 days after the second vaccine dose administered at Day 57 | Within 28 days after the second vaccine dose (administered at Day 57)
  An unsolicited AE is any untoward medical occurrence (an unfavourable/unintended sign - including an abnormal laboratory finding), symptom, or disease (new or exacerbated) in a clinical study participant that is temporally associated with the study intervention, whether or not considered related to the study intervention and that was not included in a list of solicited events using a Participant Diary.
Percentage of participants reporting medically attended AEs (MAEs) | From Day 1 up to study end at Day 421
  A MAE is an unsolicited AE for which the participants received medical attention defined as hospitalization, or an otherwise unscheduled visit to or from medical personnel for any reason, including emergency room visits.
Percentage of participants reporting serious adverse events (SAEs) | From Day 1 up to study end at Day 421
  An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study patient or results in abnormal pregnancy outcomes.
Percentage of participants reporting potential immune-mediated diseases (pIMDs) | From Day 1 up to study end at Day 421
  PIMDs are a subset of adverse events of special interest (AESIs) that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Percentage of participants reporting potential orolabial HSV-1 recurrence | From Day 1 up to study end at Day 421
  Potential orolabial HSV-1 recurrence represents a subset of adverse events of special interest (AESIs).
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at pre-vaccination (Day 1) | At pre-vaccination (Day 1)
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. In the absence of a diagnosis, abnormal laboratory findings assessments (e.g., Grade 2 or higher abnormal haematological and biochemical parameters) or other abnormal results the investigator considers clinically significant are recorded as an AE or SAE, if they meet the definition of an AE or SAE.
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at Day 2 | At Day 2
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. In the absence of a diagnosis, abnormal laboratory findings assessments (e.g., Grade 2 or higher abnormal haematological and biochemical parameters) or other abnormal results the investigator considers clinically significant are recorded as an AE or SAE, if they meet the definition of an AE or SAE.
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at Day 8 | At Day 8
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. In the absence of a diagnosis, abnormal laboratory findings assessments (e.g., Grade 2 or higher abnormal haematological and biochemical parameters) or other abnormal results the investigator considers clinically significant are recorded as an AE or SAE, if they meet the definition of an AE or SAE.
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at Day 57 | At Day 57
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. In the absence of a diagnosis, abnormal laboratory findings assessments (e.g., Grade 2 or higher abnormal haematological and biochemical parameters) or other abnormal results the investigator considers clinically significant are recorded as an AE or SAE, if they meet the definition of an AE or SAE.
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at Day 58 | At Day 58
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. In the absence of a diagnosis, abnormal laboratory findings assessments (e.g., Grade 2 or higher abnormal haematological and biochemical parameters) or other abnormal results the investigator considers clinically significant are recorded as an AE or SAE, if they meet the definition of an AE or SAE.
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at Day 64 | At Day 64
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. In the absence of a diagnosis, abnormal laboratory findings assessments (e.g., Grade 2 or higher abnormal haematological and biochemical parameters) or other abnormal results the investigator considers clinically significant are recorded as an AE or SAE, if they meet the definition of an AE or SAE.
Percentage of participants reporting any haematological and biochemical laboratory abnormalities at Day 85 | At Day 85
  Clinically significant abnormal laboratory findings are those which are not associated with an underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition. In the absence of a diagnosis, abnormal laboratory findings assessments (e.g., Grade 2 or higher abnormal haematological and biochemical parameters) or other abnormal results the investigator considers clinically significant are recorded as an AE or SAE, if they meet the definition of an AE or SAE.

SECONDARY OUTCOMES:
Anti-vaccine antibody concentrations | At pre-vaccination (Day 1), Day 29, Day 57, Day 85, Day 239 and Day 421
  Antibody concentrations determined by Enzyme Linked Immunosorbent Assay (ELISA) are presented as GMCs and expressed in ELISA unit per milliliter (EU/mL).
Percentage of seropositive participants for anti-vaccine antibodies | At pre-vaccination (Day 1), Day 29, Day 57, Day 85, Day 239 and Day 421
  The percentage of seropositive participants for anti-vaccine antibodies (i.e. participants with anti-vaccine antibody concentrations above the predefined threshold, as assessed by ELISA) is reported.
Frequency of antigen specific Cluster of Differentiation (CD)4+ T-cells expressing at least two activation markers | At pre-vaccination (Day 1), Day 29, Day 57, Day 85, Day 239 and Day 421
  Frequency of antigen-specific CD4+ T-cells is expressed as antigen-specific CD4+ T-cells per million peripheral blood mononuclear cells (antigen-specific CD4+ T-cells/million PBMCs), as assessed by cytokine flow cytometry. Among the activation markers expressed are interleukin-2/13/17 (IL-2, IL-13, IL-17), cluster of 40 ligand (CD40L), 4-1BB, tumour necrosis factor alpha (TNF-α) and interferon gamma (IFN-γ).
Frequency of antigen-specific CD8+ T-cells expressing at least two activation markers | At pre-vaccination (Day 1), Day 29, Day 57, Day 85, Day 239 and Day 421
  Frequency of antigen-specific CD8+ T-cells is expressed as antigen-specific CD8+ T-cells/million PBMCs. Among the activation markers expressed are interleukin-2/13/17 (IL-2, IL-13, IL-17), cluster of 40 ligand (CD40L), 4-1BB, tumour necrosis factor alpha (TNF-α) and interferon gamma (IFN-γ).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Rochester, New York

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.